CLINICAL TRIAL: NCT05174403
Title: Imaging Biomarkers in Spastic Paraplegia Type 5
Acronym: SPIMA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200944; IDRCB (Other: 2020-A01564-35)
Record Dates: First submitted 2020-09-14; First posted 2021-12-30 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Spastic Paraplegia Type 5A, Recessive
Keywords: spastic paraplegia; metabolism; magnetic resonance imaging; Expanded Disability Status Scale (EDSS); brain; spine
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Paraplegia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SPG5 patients: Adult SPG5 patients with diagnostic confirmed by the identification of two mutations in the CYP7B1 gene
  Interventions: Other: Cerebral and spinal cord magnetic resonance imaging

INTERVENTIONS:
Other: Cerebral and spinal cord magnetic resonance imaging — Cerebral and spinal cord magnetic resonance imaging (without injection of contrast medium).
  Patient's data will be compared to calibrated data from the commercially available medical software Brain Quant (licence BT-BQ-001-START, market CAIH, CE12331).

SUMMARY:
This is a research study aiming to identify imaging biomarkers in patients diagnosed with spastic paraplegia type 5 (SPG5)

DETAILED DESCRIPTION:
"The aim of this study is to identify robust and reliable imaging biomarkers of disease by using novel macrostructural (volumetry), microstructural (fiber tractography) and spectroscopy (metabolites) methods to calculate SPG5 patients biometrics using a commercially available medical software Brain Quant (licence BT-BQ-001-START, market CAIH, CE12331), an approach with a larger effect size than conventional methods."

This study will recruit 10 SPG5 patients. Each participant will be invited to a one-day session during which a clinical examination will performed and an EDSS score will be assigned, followed by a brain and a spine MRI/MRS examination.

Clinical implications: This study will define biomarkers that can be quantified in SPG5 patients and that could be used as read-outs to assay therapeutic effects in clinical trials focused on SPG5 patients

ELIGIBILITY:
Inclusion criteria

* At least 18 years of age
* Signature of the informed consent
* Covered by social security
* SPG5 patients identified with two mutations in the CYP7B1 gene

Exclusion criteria

* Contra-indications to MRI (claustrophobia, metallic or material implants)
* Additional psychiatric or neurological conditions / additional major comorbidities
* History of severe head injury
* Participation in another trial (except observational trial)
* Pregnancy and breastfeeding
* Inability to understand information about the protocol
* Persons under AME
* Persons deprived of their liberty by judicial or administrative decision
* Adult subject under legal protection or unable to consent
* Unwillingness to be informed in case of abnormal MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SPG5 is an Hereditary spastic paraparesis (HSP) with a frequency up to 8% of HSP families. Age at onset shows both an interfamilial and intrafamilial variability, with a range from early childhood to the 5th decade of life. Most SPG5 patients show a slowly progressive pure form.
  All carriers of SPG5 will be recruited in La Pitié-Salpêtrière Hospital (Paris) among the patients of the National Reference Centre of Rare Diseases. Initially, patients benefitted from genetic analyses (Sanger analysis or next generation sequencing panel dedicated to hereditary spastic paraplegia genes). As far as possible, cohort of SPG5 patients will be the same as the population involved in the previous clinical trial (SPA-M, NCT02314208).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Changes in the cross-sectional area in the spine of SPG5 patients | 1 day
  An MRI analysis will be performed at the level of the spinal cord of SPG5. This analysis will quantify the cross-sectional area, in pixel, of each vertebra in each imaged individual, using the commercially available medical software Brain Quant (licence BT-BQ-001-START, market CAIH, CE12331)

SECONDARY OUTCOMES:
Changes in the cross-sectional area of the segmented white matter and gray matter in the spine of SPG5 patients | 1 day
  An MRI analysis will be performed at the level of the spinal cord SPG5 patients. This analysis will quantify the cross-sectional area, in pixel2, of the segmented white matter and gray matter in each imaged individual.
Changes in the diffusion tensor imaging (DTI) of the spine in SPG5 patients | 1 day
  An MRI analysis will be performed at the level of the spinal cord of and SPG5 patients. This analysis will allow the quantification of fraction anisotropy (FA) and radial diffusivity (RD) in different regions of the spine
Changes in metabolic profiles in the spine of SPG5 patients | 1 day
  A combined MRI/MRS analysis will be performed at the level of the spinal cord of SPG5 patients. This analysis will allow to quantify in parts per million (ppm) the ratios of the following metabolites in the spine: N-acetylaspartate, myo-inositol, choline and creatine.
Changes in brain volume brain in SPG5 patients | 1 day
  An MRI analysis will be performed at the level of brain of SPG5 patients. This analysis will allow the quantification in voxels of brain volume.
Changes in the diffusion tensor imaging (DTI) in the brain of SPAG5 patients | 1 day
  An MRI analysis will be performed at the level of the brain of SPG5 patients. This analysis will allow the quantification of FA and RD in different regions of the brain.
Validation of correlation between Expanded Disability Status Scale (EDSS) score severity and severity of morphological and/or metabolic changes | 1 day
  An EDSS score will be assigned to each participant after clinical evaluation. Each participant's biomarker severity scores will be compared to his respective EDSS score and determine whether EDSS severity score correlates with biomarker severity.
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
  EDSS steps 1.0 to 4.5 refer to people who are able to walk without any aid and is based on measures of impairment in eight functional systems (FS).
  EDSS steps 5.0 to 9.5 are defined by the impairment to walking.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny MOCHEL, MD, PhD, Principal Investigator — Sorbonne Universités - Université Pierre et Marie Curie
Locations (1):
- APHP - Pitié Salpetriere Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided